CLINICAL TRIAL: NCT00666523
Title: Randomized Double-Blind Study of Food Supplement Phytalgic on Symptoms of Osteoarthritis
Brief Title: Effect of Phytalgic in Osteoarthritis (OA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université Victor Segalen Bordeaux 2 (Other)
Collaborators: laboratoire Phythea, France (Unknown)
Responsible Party: Alain Jacquet, Dept of pharmacology, CHU Bordeaux
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PhytalgicOA
Record Dates: First submitted 2008-04-23; First posted 2008-04-25 (Estimated); Last update posted 2008-04-25 (Estimated); Status verified 2008-04

CONDITIONS: Osteoarthritis
Keywords: osteoarthritis, knee or hip
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Dietary Supplement: phytalgic
- 2 (Placebo Comparator)
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: phytalgic — 3/day
  Arms: 1
Dietary Supplement: placebo — 3/Day
  Arms: 2

SUMMARY:
The objective of the study is to test the effects of a herbal supplement, Phytalgic, on the symptoms of osteoarthritis of the knee or hip, in patients with OA using NSAIDs or analgesics on a regular basis.

ELIGIBILITY:
Inclusion Criteria:

* knee or hip osteoarthritis
* regular NSAIDs/analgesic treatment
* signed inform consent

Exclusion Criteria:

* incapacity to understand study
* irregular NSAID treatment

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2007-01; Primary Completion 2008-01 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
use of NSAIDs or analgesics | 3 months

SECONDARY OUTCOMES:
WOMAC function scale | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Moore, MD, PhD, Study Director — University of Bordeaux
Locations (1):
- Dept of Pharmacology, U-Bordeaux2, BP36, Bordeaux, France

REFERENCES:
- [Derived] Jacquet A, Girodet PO, Pariente A, Forest K, Mallet L, Moore N. Phytalgic, a food supplement, vs placebo in patients with osteoarthritis of the knee or hip: a randomised double-blind placebo-controlled clinical trial. Arthritis Res Ther. 2009;11(6):R192. doi: 10.1186/ar2891. Epub 2009 Dec 16. PMID 20015358